CLINICAL TRIAL: NCT04267978
Title: Open-label Prospective Study of Recombinant Human Endostatin Combined with Cytotoxic Chemotherapy Regimen in the Treatment of Recurrent Gliomas
Brief Title: Study of Recombinant Human Endostatin Combined with Temozolomide and Irinotecan in Recurrent Gliomas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Sanbo Brain Hospital (Other)
Responsible Party: Principal Investigator, Junping Zhang, Chief physician, Beijing Sanbo Brain Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBNK-YJ-2019-006-02
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Glioblastoma, Recurrent; Lower Grade Glioma, Recurrent
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — Endostatins

STUDY DESIGN:
Intervention Model Description: glioblastoma, lower-grade glioma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- glioblastoma (Experimental)
  Interventions: Drug: recombinant human endostatin,temozolomide,irinotecan
- lower-grade glioma (Experimental)
  Interventions: Drug: recombinant human endostatin,temozolomide,irinotecan

INTERVENTIONS:
Drug: recombinant human endostatin,temozolomide,irinotecan — Temozolomide was given orally 200mg/m2 for 5 days in each cycle. Day 1 TMZ was administered 3-6 hours prior to irinotecan.
  Irinotecan was administrated 125mg/m2 on day 1 and day 15. Recombinant human endostatin was administrated 15mg/d, daily for 14 days. One treatment cycle was defined as 28 days (4 weeks), even if treatment is held mid-cycle for toxicity.
  Treatment was continued until disease progression, patient withdrawal, or unacceptable toxicity.
  The maximum number of treatment cycles was 12. After 12 cycles of treatment, if the investigator judges that the subject may continue to benefit from the regimen, the duration of treatment may be extended with the subject's consent.

SUMMARY:
Almost all gliomas relapse. After temozolomide rechallenge or combination with irinotecan, the progression-free survival rate at 6 months (PFS-6%) of recurrent glioblastoma was about 21%. After treatment with irinotecan-based chemotherapy regimen, the PFS-6% of recurrent lower-grade gliomas was 40%. The optimal chemotherapeutics of recurrent gliomas has yet to be determined.

Anti-angiogenesis is a promising therapeutic strategy. Vascular endothelial growth factor-A (VEGF) is the primary driver of angiogenesis in tumors. Bevacizumab, a humanized monoclonal antibody directed against VEGF, is the prototypical anti-angiogenic drug and received accelerated approval of the United States Food and Drug Administration (FDA) for the treatment of recurrent glioblastoma. Bevacizumab inproved the PFS-6% (36%), but had no effect on the overall survival (OS) (9.2 months). Moreover, the effects of bevacizumab are transient and most patients' tumors progress just after a median time of 3-5 months. Recombinant human endostatin (rh-ES) is an endogenous broad-spectrum angiogenesis inhibitor that has been shown to significantly improve therapeutic efficacy when combining with conventional chemotherapy agents in non-small-cell lung cancer, breast cancer and melanoma.

In our previous study, we retrospectively analyzed the effect and toxicity of rh-ES when combined with temozolomide and irinotecan on adult recurrent disseminated glioblastoma. After combined treatment, PFS-6% was 23.3%; the median PFS and OS were 3.2 and 6.9 months, respectively, which were promising compared with that in other studies. Once patients get radiographic remission in a short time (4 months), they may get a long PFS.The combined regimen did not reduce the sensitivity of tumor to bevacizumab. After tumor progression from the combined chemotherapy, bevacizumab usage could help to prolong the survival time (5.1 months versus 2.4 months). Moreover, the toxicities of the combination therapy in this study were manageable.

On the basis of prior clinical experience, we carry out this prospective trial to confirm the efficacy and safety of the combination of rh-ES, temozolomide and irinotecan in patients with recurrent gliomas.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤70;
2. Histopathologically-confirmed, supratentorial GBM or lower-grade gliomas (such as oligodendroglioma, astrocytoma, oligoastrocytoma, anaplastic astrocytoma, anaplastic oligodendroglioma or anaplastic oligoastrocytoma);
3. Recurrence is pathologically confirmed by another biopsy or surgery, which should have been completed at least 2 weeks before enrollment, or confirmed by the MRI according to RANO criteria, at least one bi-dimensionally measurable contrast-enhancing target lesion, with one diameter at least 10 mm, visible on two or more axial slices 5mm apart;
4. Received standard chemoradiotherapy and at least one cycle of chemotherapy after primary diagnosis;
5. The time intervals between the last radiotherapy and enrollment are at least 3 months;
6. The interval form the last chemotherapy to the study enrollment was at least one interval of chemotherapy with recover from the related toxic effects (except for hair loss and pigmentation);
7. Karnofsky Performance Status ≥ 60;
8. If the patient is on glucocorticoid therapy, hormone dosage should be stable or decreased at least 5 days before baseline MRI;
9. If the patient is receiving enzyme-inducing antiepileptic drugs (EIAEDs), the drugs should be replaced with non-EIAEDs for at least 1 weeks away from enrollment;
10. Estimated survival of at least 12 weeks;
11. Participants must have adequate organ function as defined by the following criteria (within 7 days before treatment):

    1. Hematology (No transfusion within 14 days):

       * Hemoglobin(HB)≥90g/L;

         * Absolute neutrophil count (ANC)≥1.5×109/L;

           * Platelet (PLT)≥80×109/L.
    2. Chemistry:

       * Serum bilirubin ≤ 1.5×upper limit of normal (ULN)

         * ALT and AST≤2.5ULN；

           * Serum creatinine ≤1.5ULN or creatinine clearance rate(CCr)≥60ml/min；
    3. ECG: heart rate in the normal range (55-100beats/min), normal or slightly prolonged QT interval (QTc<480ms), normal or low T wave, normal or non-specific ST segment changes.
12. Both men and women at the gestational age must agree to take adequate contraceptive measures throughout the study period.
13. Participants volunteered to participate in the study and signed an informed consent form (ICF)

Exclusion Criteria:

1. MRI examination is not available (such as pacemaker, metal denture);
2. Receiving any other investigational agent.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the drugs used in this study.
4. Patients who have received organ transplants.
5. Patients with HIV or Treponema pallidum infection.
6. Severe heart disease; ECG shows T wave inversion or elevation or ST segment specific changes.
7. Having factors that affect oral drug absorption, such as vomiting, diarrhea and intestinal obstruction
8. There were clinically significant bleeding symptoms or clear bleeding tendency in the first 3 months before enrollment, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, gastrointestinal perforation, baseline fecal occult blood ++ and above, intracranial or intracranial hemorrhage, or vasculitis;
9. Arteriovenous thrombosis events occurred within 6 months before enrollment, such as cerebrovascular accidents (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.;
10. Having bleeding disorder and are being treated with thrombolytic or anticoagulant drugs.
11. Other conditions considered inappropriate by the researcher for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2020-02-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival rate at 6 months | up to 4 years
  the percentage of participants who remained progression free at 6 months after treatment initiation.

SECONDARY OUTCOMES:
objective response rate | up to 4 years
  the percentage of patients who achieved confirmed complete response or partial response according to the Response Assessment in Neuro-Oncology (RANO) criteria.
Progression-free survival | up to 4 years
  the time interval from treatment initiation to disease progression or death, whichever occurs first.
Overall survival | up to 4 years
  the time interval from treatment initiation to death from any cause.
Safety data | up to 4 years
  Frequency and severity of adverse effects as defined by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Jun-ping Zhang, Principal Investigator — Beijing Sanbo Brain Hospital
Locations (1):
- Beijing Sanbo Brain Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No